CLINICAL TRIAL: NCT04139941
Title: Prospective Diagnostic Accuracy Study of Rapid Diagnostic Tests (RDTs) Detecting Antibodies Against Hepatitis C Virus (HCV) in Freshly Collected Whole Blood, Plasma and Serum
Brief Title: Evaluation Study of HCV RDTs in Fresh Samples
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: 8162-2/2
Record Dates: First submitted 2019-10-07; First posted 2019-10-25 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Left-over and unused back up samples of plasma and serum will be stored at a bio-repository
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with known or unknown HCV status
  Interventions: Diagnostic Test: Test for HCV antibodies with an RDT

INTERVENTIONS:
Diagnostic Test: Test for HCV antibodies with an RDT — Fingerstick whole blood, plasma and serum of each participant is tested with three investigational HCV RDTs and one reference HCV RDT. Plasma is also used for testing with the composite reference standard, HCV viral load and genotyping. All participants are also tested for HIV with an HIV RDT.

SUMMARY:
This study evaluates the sensitivity and specificity performance of three Hepatitis C Virus (HCV) rapid diagnostic tests (RDTs) in freshly collected fingerstick whole blood, as well as serum and plasma (Premier Medical Corporation First Response HCV RDT; Beijing Wantai HCV RDT; AccessBio Care Start HCV under development). Performance is compared to the SD Bioline HCV RDT, as well as a composite reference standard, consisting of two enzyme Immunoassay and a line immunoassay.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is a major public health burden, with an estimated 71 million patients being infected globally. If undiagnosed, HCV infection can lead to severe liver damage, including hepatocellular carcinoma (HCC). The World Health Organization (WHO) recently set a target to eliminate HCV by 2030. The first critical step in reaching this target is to accurately identify people infected with HCV. Globally, significant gaps remain in diagnosis of HCV, with four out of five people infected still unaware of their status, largely due to lack of access to testing services.

In resource-limited settings (RLS), laboratory-based testing remains a mainstay for HCV screening and confirmatory testing. Such laboratory-based assays rely on transportation of temperature-sensitive samples from clinic sites to centralized laboratories, high-tech equipment and highly skilled laboratory technicians, limiting the scope of access to testing and resulting in long turn-around times for results. In recent years, new technologies have been developed to decentralize HCV screening and confirmatory testing using point-of-care (POC) assays to overcome these barriers and improve patient outcomes.

Rapid diagnostic tests (RDT) for screening for HCV are affordable, accurate, easy to use by healthcare workers, and robust in field settings. Although a number of HCV RDTs are on the market, currently only two have received WHO pre-qualification (PQ) status, demonstrating their accuracy and reliability for use in the field in RLS. Data on a number of other RDTs indicate their suitability for use. More data is needed, however, in field settings for these HCV RDTs, to demonstrate their accuracy and quality in end-user studies and to provide evidence for WHO PQ approval.

Based on the results of a recent FIND laboratory evaluation assessing the performance of 13 HCV RDTs using archived plasma samples, we have selected three candidate HCV RDTs ("study RDTs") for further evaluation in field settings (e.g. primary healthcare facilities). The performance of these RDTs measured in frozen plasma specimens indicated that they have a high potential to meet WHO PQ performance criteria in freshly collected samples. In addition, the manufacturers each demonstrate evidence of engagement to pursue both CE-mark status and the WHO PQ process, showing commitment to delivering quality-assured tests to the market.

The data generated during this study will be used to inform national and international stakeholders on HCV RDT performance in field settings and shared with manufacturers to support the evidence package for WHO PQ and/or CE-marking.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Known or unknown HCV serology
* No history of past or present HCV treatment
* Willing to undergo the information and consenting procedure and subsequently have enough time to participate in the study
* Willing to provide 13 ml venepuncture blood sample and a minimum of four whole blood fingerstick samples
* Willing to perform an HIV test
* Individuals can already be registered at the local site or register for the first time when enrolling in the study

Exclusion Criteria:

* Participants not able to consent themselves (incapable)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * General population
  * HCV high-risk individuals
Sampling Method: Probability Sample
Enrollment: 1540 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of HCV RDTs compared to a composite reference standard | through study completion, on average 1 year
  1.1 Point estimates of sensitivity, specificity, positive and negative predicative values (with 95% confidence intervals) and Cohen's Kappa Coefficient (κ) of inter-rater agreement for each RDT, using a combination of two EIAs (Enzyme Immunoassay) and an LIA (Line immunoassay) as a composite reference standard for the detection of anti-HCV antibodies in fingerstick whole blood, EDTA plasma and serum.

SECONDARY OUTCOMES:
Sensitivity and specificity of HCV RDTs compared to an HCV RDT pre-qualified by WHO as reference standard | through study completion, on average 1 year
  2.1 Point estimates of sensitivity, specificity, positive and negative predicative values (with 95% confidence intervals) and Cohen's Kappa Coefficient (κ) of inter-rater agreement for each RDT, using the WHO-PQ RDT as reference standard for the detection of anti-HCV antibodies in fingerstick whole blood, EDTA plasma and serum
Operational characteristics | through study completion, on average 1 year
  2.2 Operational characteristics and usability of study RDTs:
  - Rate of invalid test results /errors: Percentage of invalid test results/errors by RDT, site and error type
Operational characteristics | through study completion, on average 1 year
  Operational characteristics and usability of study RDTs:
  - Technical appraisal rating on kit instructions, labelling and test conduct, on a Likert scale

CONTACTS AND LOCATIONS:
Locations (2):
- Sihanouk Hospital Centre of Hope, Phnom Penh, Cambodia
- National Center for Disease Control & Public Health/Lugar Center, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be shared with the manufacturers who's RDTs are being evaluated
Supporting Information: CSR
Time Frame: end of study